CLINICAL TRIAL: NCT00741806
Title: Randomized, Double-blind, Placebo-controlled, Phase I Dose-escalation Study of Single Dose GHB04L1 in Healthy Adults
Brief Title: Dose-escalation Study of Single Dose GHB04L1 in Healthy Adults
Acronym: GHB-CS03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVIR Green Hills Biotechnology AG (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: AVIR Green Hills Biotechnology AG, AVIR Green Hills Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GHB-CS03; EudraCT 2007-003219-29
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: vaccination; avian
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GHB04L1 (Experimental): Single dose, dose escalation
  Interventions: Biological: GHB04L1
- SPGN buffer (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GHB04L1 — single dose intranasal administration of GHB04L1
  Other Names: A/Vietnam/1203/04 (H5N1)-ΔNS1 virus reassortant
  Arms: GHB04L1
Other: Placebo — SPGN buffer
  Arms: SPGN buffer

SUMMARY:
It is the hypothesis of this study that intranasal vaccination with a single dose of GHB04L1 is safe and induces an immune response against influenza A H5N1. This hypothesis will be tested in a randomized, double-blind, placebo-controlled, Phase I dose-escalation study assessing the safety and tolerability of single dose administration of GHB04L1 in healthy adults. Furthermore, the local and systemic immune response as well as the pharmacokinetic properties of a single dose of GHB04L1 will be studied as secondary objectives. GHB04L1 will be escalated according to a fixed dose escalation scheme comprising three dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18-50 years
* Seronegative for H5N1
* Seronegative for H1N1 (with antibody titers ≤1:20)
* Written informed consent to participate in this study

Exclusion Criteria:

* Acute febrile illness
* Signs of acute or chronic upper or lower tract respiratory illnesses
* History of severe atopy
* Seasonal influenza vaccination from 2006/2007 onwards and/or pandemic influenza vaccination against H5N1
* Known increased tendency of nose bleeding
* Volunteers with clinically relevant abnormal paranasal anatomy
* Volunteers with clinically relevant abnormal laboratory values
* Simultaneous treatment with immunosuppressive drugs
* Clinically relevant history of renal, hepatic, GI, cardiovascular,haematological, skin, endocrine, neurological or immunological diseases
* History of leukaemia or cancer
* HIV or Hepatitis B or C seropositivity
* Volunteers who underwent rhino or sinus surgery, or surgery of another traumatic injury of the nose within 30 days prior to application of study medication
* Volunteers who have received antiviral drugs, treatment with immunoglobulins or blood transfusions, or an investigational drug within four weeks prior to study medication application
* Volunteers who have received anti-inflammatory drugs 2 days prior to study medication application
* Volunteers who are not likely to cope with the requirements of the study or with a significant physical or mental condition that may interfere with the completion of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of GHB04L1 administered as single dose intranasal aerosol for vaccination against influenza A (H5N1) virus. | study medication administration until 30 days after end of study

SECONDARY OUTCOMES:
To assess local immune response, systemic immune response and pharmacokinetics (shedding) of a single dose of GHB04L1 aerosol administered intranasally. | day1 until day 29

CONTACTS AND LOCATIONS:
Overall Officials: Volker Wacheck, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept of Clinical Pharmacology, Medical University Vienna, Vienna, Austria